CLINICAL TRIAL: NCT00841269
Title: Oral Administration of Uridine for Treatment of Bipolar Depression in Adolescents: A Magnetic Resonance Spectroscopy Study
Brief Title: Oral Uridine for Treatment of Bipolar Depression in Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Douglas Kondo, MD, MD, University of Utah
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 28455; 5R01MH058681-06 (NIH)
Record Dates: First submitted 2009-02-09; First posted 2009-02-11 (Estimated); Results first posted 2015-01-08 (Estimated); Last update posted 2018-03-26 (Actual); Status verified 2018-02

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Manic Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — Uridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Uridine (Experimental): Uridine 500 mg by mouth twice daily for 6 weeks
  Interventions: Drug: Uridine
- Healthy Comparison (No Intervention): Healthy comparison participants were seen for baseline and week 6 MRI scans. No treatment was administered to participants enrolled as healthy comparisons.

INTERVENTIONS:
Drug: Uridine — Uridine 500 mg by mouth twice per day for 6 weeks
  Arms: Uridine

SUMMARY:
The purpose of the study is to see if the investigational medication uridine reduces depression symptoms in adolescents with bipolar disorder. Uridine is a naturally occurring chemical that is made by the human liver. Uridine is part of a family of compounds called pyrimidines, and is normally involved in many of the body's processes such as the use of energy by cells. Uridine is considered experimental, because it has not been approved by the U.S. Food and Drug Administration (FDA) to treat bipolar depression in adolescents. The study will use standard methods of assessing adolescent's mood, such as rating scales and questionnaires. In addition, the study will use Magnetic Resonance Imaging Spectroscopy (MRI/MRS) brain scans to see if levels of certain chemicals in the brain change when adolescents are treated with uridine. These scans use a magnet to create images of the brain, and do not expose patients to radiation.

DETAILED DESCRIPTION:
This is an open-label study of the investigational drug uridine in the treatment of adolescents with depression with bipolar disorder. Uridine has shown positive results in a Phase II study of bipolar disorder in adults (http://clinicaltrials.gov/ct2/show/NCT00322764). This study will enroll 30 depressed adolescent participants who meet DSM-IV-TR criteria for bipolar disorder type I, type II or bipolar disorder not otherwise specified. Participants who are currently taking psychotropic medication(s) will continue on their current regimen, with uridine added as adjunctive therapy. Participants who are untreated will be informed of the alternatives to study participation. This will include informing the parent(s) or guardian(s) that Lithium, Risperdal and Abilify are FDA-approved treatments for adolescent bipolar disorder that would be available to their child in community care.

The study has three objectives: 1) To use Magnetic Resonance Spectroscopy (MRS) brain imaging to measure levels of beta-nucleoside triphosphate (b-NTP) in the anterior cingulate cortex of 30 adolescents with bipolar disorder, before-and-after 6 weeks of treatment with the investigational drug uridine; 2) To measure the antidepressant response to uridine in the 30 participants with the Children's Depression Rating Scale (CDRS); and 3) To acquire structural Magnetic Resonance Imaging (MRI) data in the 30 participants with bipolar disorder and the 30 healthy controls, to establish regionally-specific structure/neurochemical relationships.

Adolescent participants with bipolar disorder will be treated with uridine 500mg twice daily for six weeks. The primary clinical outcome measure is the Children's Depression Rating Scale (CDRS), with response defined as a 30% reduction in CDRS score. In addition to this standardized clinical assessment, participants will undergo magnetic resonance imaging and magnetic resonance spectroscopy (MRI/MRS) brain scans at baseline, and after six weeks of treatment with uridine. This novel approach is designed to explore objectively measurable biomarkers of illness and treatment response in pediatric bipolar disorder. The investigators hypothesize that participants whose depression responds to uridine will demonstrate an increased concentration of beta-nucleoside triphosphate (b-NTP) in the anterior cingulate cortex. This would support the hypothesis that depressive states are associated with abnormalities in brain energy metabolism.

As a neuroimaging comparison group for the participants with bipolar disorder, 30 healthy adolescent controls with no history of psychiatric illness will be recruited for MRI/MRS scanning only. The investigators hypothesize that controls will have higher levels of b-NTP in the anterior cingulate cortex than participants with depression associated with bipolar disorder, further supporting a connection between brain bioenergetics and depression.

ELIGIBILITY:
Selection of Participants with Bipolar Disorder:

Inclusion Criteria:

* Participants must meet DSM-IV-TR (American Psychiatric Association, 2000) criteria for Bipolar Disorder Type I, Type II, or Not Otherwise Specified (NOS) with current mood state depressed for > 2 weeks
* Participants must be between the age of 13 and 18 years
* Participants who enter the study on psychotropic medications must be on a regimen that has been stable for > 2 weeks at the time of study entry
* Participants must be able to give informed consent or assent, and parent(s)/guardian(s) must be able to give informed permission for study participation

Exclusion Criteria:

* Adolescents with an unstable co-morbid medical, neurological, or psychiatric disorder
* Pregnant females, nursing mothers, or females of childbearing potential who are unable or unwilling to practice contraception during the study
* Participants with high risk of suicidal behaviors, homicidal behaviors, or self-harm
* Participants who in the opinion of the investigator are unlikely to be able to comply with the study protocol
* Participants who meet DSM-IV-TR criteria for current substance abuse or substance dependence, with the exception of nicotine abuse or dependence
* Participants for whom the MRI/MRS scans are contraindicated, such as children with ferromagnetic implants or claustrophobia
* Participants whose mood state is manic
* Documented or suspected history of mental retardation (IQ<70)
* Positive urine drug screen for cocaine or amphetamines
* Known hypersensitivity to uridine

Selection of Healthy Volunteers:

Inclusion Criteria:

* Participants must be between the ages of 13 and 18 years
* Participants must not meet DSM-IV-TR diagnostic criteria for a mental disorder or substance abuse
* Participants must be able to give informed consent or assent and parents/guardians must be able to give informed permission for participation

Exclusion Criteria:

* Clinically significant medical, neurological, psychiatric or substance abuse disorder
* Pregnant subjects, due to the unknown effects of MRI/MRS scans on a fetus. In addition, women of childbearing potential who are unable or unwilling to practice contraception during the study will be excluded. Female participants who are of child-bearing potential must have a negative urine pregnancy test before each MRI/MRS scan.
* Participants with a contraindication to MRI/MRS scanning, such as a metallic implant
* Patients unable to comply with the protocol

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2009-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas G Kondo, M.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah School of Medicine, Salt Lake City, Utah, United States

REFERENCES:
- [Result] Kondo DG, Sung YH, Hellem TL, Delmastro KK, Jeong EK, Kim N, Shi X, Renshaw PF. Open-label uridine for treatment of depressed adolescents with bipolar disorder. J Child Adolesc Psychopharmacol. 2011 Apr;21(2):171-5. doi: 10.1089/cap.2010.0054. Epub 2011 Apr 12. PMID 21486171
- See also: UtahBrain.org — http://UtahBrain.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via clinician referrals and IRB-approved recruitment materials and advertising.
Groups:
- Open Label Uridine Treatment: Participants received fixed-dose uridine 500 mg twice daily for 6 weeks. At each treatment visit, the following rating scales were administered: The CDRS-R, YMRS, and the Columbia-Suicide Severity Rating Scale (C-SSRS)
- Healthy Comparison: Participants assigned to this group were seen for two scan visits (baseline and week 6). Healthy comparison participants received no intervention.
Period: Overall Study
Arm/Group | Open Label Uridine Treatment | Healthy Comparison
Started | 20 | 22
Completed | 12 | 13
Not Completed | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Open Label Uridine Treatment: All participants were Caucasian. There were 5 female participants and 2 male participants.
- Healthy Comparison: Participants assigned to this group were seen only at baseline and received no intervention.
- Total: Total of all reporting groups
Arm/Group | Open Label Uridine Treatment | Healthy Comparison | Total
Number analyzed (Participants) | 20 | 22 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 18 | 38
  Between 18 and 65 years | 0 | 4 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.05 (1.50) | 15.67 (1.84) | 15.83 (1.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 11 | 13 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 20 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 22 | 42

OUTCOME MEASURES:

1. Primary Outcome: Mean Scores in Children's Depression Rating Scale (CDRS-R), Assessed Before and After 6 Week Uridine Treatment
Description: The CDRS-R is a 17-item scale, with items rated for severity on a 5 point scale for 3 items and on a 7 point scale for 14 items (possible total score from 17 to 113). Ratings are completed by a clinician via interviews with the child or parent. Scores ≥40 are indicative of depression, whereas scores ≤28 is often used to define remission.
Time Frame: 6 weeks
Measure: Mean (Full Range); unit: Units on a scale
Groups:
- Open Label Uridine Treatment: Participants received fixed-dose uridine 500 mg twice daily for 6 weeks.
- Healthy Comparison: Participants assigned to this group were seen for two scan visits (baseline and week 6). Healthy comparison participants received no intervention/treatment.
Arm/Group | Open Label Uridine Treatment | Healthy Comparison
Number analyzed (Participants) | 12 | 13
Units on a scale
  before treatment | 60.00 [40 to 82] | 21.29 [17 to 35]
  after 6 week Uridine treatment | 33.83 [20 to 59] | 20 [17 to 25]

2. Primary Outcome: The Primary Neuroimaging Outcome Will be Changes in Beta-NTP to TP (Total Phosphorus) Ratio in the Anterior Cingulate.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Beta-NTP/TP Ratio
Arm/Group | Open Label Uridine Treatment | Healthy Comparison
Number analyzed (Participants) | 12 | 13
Beta-NTP/TP Ratio
  Before treatment | 0.1168 (0.0157) | 0.1232 (0.0127)
  After 6 weeks treatment | 0.1193 (0.0142) | 0.1297 (0.0140)

3. Secondary Outcome: A Secondary Outcome Measure Includes a Change in Young Mania Rating Scale (YMRS) Score
Description: The Young Mania Rating Scale (YMRS) is an 11-item rating scale that evaluates manic symptoms. Total scores range from 0-60, with higher scores indicating more manic symptoms endorsed by research participants.
Time Frame: 6 weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Open Label Uridine Treatment | Healthy Comparison
Number analyzed (Participants) | 12 | 13
units on a scale
  Before treatment | 5.42 [2 to 11] | 0.7083 [0 to 6]
  After 6 weeks treatment | 3.08 [0 to 7] | 2.1818 [0 to 9]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from participants at every visit, starting after the treatment intervention was dispensed at baseline. Adverse events were assessed up to 6 weeks.
Description: Healthy comparison participants were only seen for scans at baseline and week 6. Healthy comparison participants were not exposed to any treatment intervention, therefore, adverse events were not collected.
Groups:
- Uridine 500 mg by Mouth Twice Daily for 6 Weeks: Because this was an open-label study, all participants received the investigational drug uridine.
Arm/Group | Uridine 500 mg by Mouth Twice Daily for 6 Weeks
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 6/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Uridine 500 mg by Mouth Twice Daily for 6 Weeks (N=20)
Suicidal ideation (Psychiatric disorders) | 1 (1) — A 17 year old male participant had suicide ideation that occurred 2 weeks after he completed the study and stopped the investigational drug. It was determined that this serious adverse event was expected, and not related to the study medication.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Uridine 500 mg by Mouth Twice Daily for 6 Weeks (N=20)
suicidal ideation (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (4)
Abdominal cramp, Nausea, Indigestion (Gastrointestinal disorders) | 6 (10)
Flu-like symptoms (fatigue, bronchitis, sinusitis) (General disorders) | 6 (7)
Hordeolum (Eye disorders) | 1 (1)
Back pain (General disorders) | 1 (1)
Vivid Dreams (Psychiatric disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Limited sample size and small percentage of underrepresented racial/ethnic minority participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No